CLINICAL TRIAL: NCT05173779
Title: A Single-arm Study to Evaluate the Efficacy and Safety of Left Atrial Isolation Achieved by Catheter Ablation in Patients With Persistent Atrial Fibrillation and Severe Atrial Fibrosis: a Chinese Registry Study
Brief Title: Left Atrial Isolation by Catheter Ablation in Persistent Atrial Fibrillation With Severe Atrial Fibrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Xu Liu, Professor, deputy director of cardiology department of Shanghai Chest Hospital, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAICA
Record Dates: First submitted 2021-12-14; First posted 2021-12-30 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Persistent Atrial Fibrillation; Severe atrial fibrosis; Left atrial isolation; catheter ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Left atrial isolation arm (Experimental): All the enrolled subjects will receive left atrial isolation through catheter ablation.
  Interventions: Procedure: Left atrial isolation by catheter ablation

INTERVENTIONS:
Procedure: Left atrial isolation by catheter ablation — Procedure: Right pulmonary vein circumferential isolation + anterior left atrial line (superior mitral annulus to right superior pulmonary vein via the anterior wall) + para-septal line (para-septal mitral annulus to the right inferior pulmonary vein, including right atrial components-especially in and around the proximal coronary sinus) + posterior left atrial line (superior mitral annulus to right superior pulmonary vein via the posterior wall).

SUMMARY:
This is a single-arm clinical trial evaluating the efficacy and safety of left atrial isolation achieved by catheter ablation in patients with persistent atrial fibrillation with severe atrial fibrosis.

DETAILED DESCRIPTION:
This is a single-arm clinical trial. Patients with persistent atrial fibrillation with severe atrial fibrosis are enrolled as subjects to conduct left atrial isolation by catheter ablation. Postoperative recurrence rate and other indicators are analyzed to evaluate the efficacy and safety of left atrial isolation achieved by catheter ablation in patients with persistent atrial fibrillation with severe atrial fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 80 years old
2. Persistent AF with severe atrial fibrosis and left atrial anterioposterior diameter > 50mm
3. Nonresponse or intolerance to ≥1 antiarrhythmic drug
4. CHA2DS2-VASc ≥ 3 and HAS-BLED < 3

Exclusion Criteria:

1. With uncontrolled congestive heart failure;
2. Having significant valvular disease;
3. Having moderate-to-severe pulmonary hypertension;
4. With myocardial infarction or stroke within 6 months of screening;
5. With Significant congenital heart disease;
6. Ejection fraction was <40% measured by echocardiography;
7. Allergic to contrast media;
8. Contraindication to anticoagulation medications;
9. Severe pulmonary disease e.g. restrictive pulmonary disease, chronic obstructive disease (COPD);
10. Left atrial thrombus;
11. Having any contraindication to right or left sided heart catheterization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative atrial fibrillation (AF)/atrial flutter (AFL)/atrial tachycardia (AT) recurrence rate | up to 18 months after enrollment
  AF/AFL/AT recurrence is defined as presence of documented AF/AFL/AT episodes of 30 seconds or longer duration

SECONDARY OUTCOMES:
Postoperative AF recurrence rate | up to 18 months after enrollment
  AF recurrence is defined as presence of documented AF episodes of 30 seconds or longer duration
Postoperative AFL/AT rate | up to 18 months after enrollment
  Occurrence of AFL/AT is defined as presence of documented AFL/AT episodes of 30 seconds or longer duration
Incidence of complications | up to 18 months after enrollment
  including death, atrio-esophageal fistula, cardiac tamponade/perforation, myocardial infarction, stroke/cerebrovascular accident, thromboembolism, diaphragmatic paralysis, pneumothorax, pleural effusion, heart block, pulmonary vein stenosis, pulmonary edema, left atrial thrombus, pericarditis and major vascular access complication or bleeding
Changes in the diameter of the left atrium and the left ventricular ejection fraction | up to 18 months after enrollment